CLINICAL TRIAL: NCT03067012
Title: Nutritional Safety and Metabolic Benefits of Oncometabolic Surgery (Long Limb Uncut Roux-en Y Gastrojejunostomy) for Obese Gastric Cancer
Brief Title: Nutritional Safety and Metabolic Benefits of Oncometabolic Surgery for Obese Gastric Cancer Patients
Acronym: ONCOMETAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Young Suk Park, Clinical Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH010
Record Dates: First submitted 2017-02-23; First posted 2017-03-01 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Oncology; Metabolic Disease; Gastric Cancer
Keywords: Oncometabolic surgery; Long limb uncut Roux-en-Y gastrojejunostomy; Obesity; Diabetes; Early gastric cancer
MeSH Terms: conditions — Neoplasms; Metabolic Diseases; Stomach Neoplasms; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncometabolic reconstruction (Experimental): Patients undergoing oncometablic surgery
  Interventions: Other: Oncometabolic reconstruction

INTERVENTIONS:
Other: Oncometabolic reconstruction — The length of biliopancreatic limb is 50cm and the length of Roux limb is 100cm. (long limb uncut Roux-en-Y gastrojejunostomy) These limbs are longer than the conventional uncut Roux-en-Y reconstruction for gastric cancer patients.

SUMMARY:
The metabolic effect of oncometabolic surgery (long limb Roux-en Y reconstruction) for early gastric cancer patients has been revealed in a few pilot studies. However, the nutritional safety has not been dealt with in previous literatures. This is a prospective pilot study for evaluating the nutritional safety and metabolic benefits of oncometabolic surgery for obese early gastric cancer patients.

DETAILED DESCRIPTION:
We performed long limb uncut Roux-en Y gastrojejunostomy (uRYGJ) in 20 patients with clinical T1N0 stage and preoperative body mass index (BMI) ≥ 32.5 kg/m2 or ≥ 27.5 kg/m2 with co-morbidities between September 2015 and July 2016.

The primary endpoint was the incidence of micronutrients' deficiency (iron, folate, vitamin B12) at postoperative 1 year and secondary endpoints were anemia incidence, BMI change and remission rates of co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Lesion located on distal or mid stomach Lesion confined to submucosa (cT1b) : Early gastric cancer No evidence of metastatic enlarged lymph nodes Preoperative body mass index (BMI) ≥ 32.5 kg/m2 or ≥ 27.5 kg/m2 with co-morbidities

Exclusion Criteria:

* Being unable to understand the risks, benefits and compliance requirements of this trial Non- Korean speaker American society of anesthesiology (ASA) class IV or higher Other malignancy within 5 years.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
micronutrients' deficiency (iron, folate, vitamin B12) | postoperative 1-year
  Iron deficiency : serum ferritin < 20 μg/dL, Vitamin B12 deficiency : serum vitamin B12 < 200 pg/mL,

SECONDARY OUTCOMES:
anemia incidence | postoperative 1-year
  Iron deficiency anemia : anemia with concomitant iron deficiency, Anemia of chronic illness : anemia with serum ferritin > 20 μg/dL, Anemia from vitamin B12 deficiency : megaloblastic anemia (MCV >100 fL) with vitamin B12 deficiency
Body mass index (BMI) change | postoperative 1-year
  Preoperative BMI minus postoperative BMI
Remission rates of co-morbidities | postoperative 1-year

IPD SHARING:
Plan to Share IPD: No